CLINICAL TRIAL: NCT05782725
Title: Subclinical Hypothyroidism and Ovarian Reserve Indices in Women With Normogonadotropic Anovulation
Brief Title: Subclinical Hypothyroidism and Normogonadotropic Anovulation
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, Principal Investigator, Jagiellonian University
Other Study IDs: 1072.6120.172.2022
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Polycystic Ovary Syndrome; Hypothalamic-Pituitary-Ovarian Axis Dysfunction (Disorder)
Keywords: Polycystic ovary syndrome; Hypothalamic-Pituitary-Ovarian axis dysfunction; Ovarian reserve; Anovulation; Any-Mullerian hormone
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: PCOS and SCH
  Interventions: Other: Comparison of laboratory test results in women in the 4 study arms
- 2: PCOH without SCH
  Interventions: Other: Comparison of laboratory test results in women in the 4 study arms
- 3: HPOD and SCH
  Interventions: Other: Comparison of laboratory test results in women in the 4 study arms
- 4: HPOD without SCH
  Interventions: Other: Comparison of laboratory test results in women in the 4 study arms

INTERVENTIONS:
Other: Comparison of laboratory test results in women in the 4 study arms — Comparison of AMH, FSH, LH, estradiol, AFC/ ovarian volume on ultrasound in women in the 4 study arms

SUMMARY:
Thyroid hormones (TH) can modify the functioning of the hypothalamic-pituitary-ovarian axis, affecting the functions of granulosa cells and the development and apoptosis of preantral follicles. TH receptors are present within the oocytes, and TH and anti-thyroid antibodies (ATA) are present in the follicular fluid. Improper thyroid function can cause ovulation disorders, luteal phase failure, impaired endometrial receptivity and result in implantation failures and recurrent miscarriages. While overt hypothyroidism is treated to improve fertility, the effect of subclinical hypothyroidism (SCH) and the presence of circulating ATAs on fertility and obstetric outcomes is uncertain and data on ovarian reserve rates are conflicting. Among the causes of ovulation disorders (group II according to the WHO classification), polycystic ovary syndrome (PCOS) dominates, found in 3-15% of women of reproductive age, and the remaining group of causes is the so-called Hypothalamic-Pituitary-Ovarian Axis Dysfunction (HPOD). The exact etiology of both entities is unknown.

DETAILED DESCRIPTION:
Purpose of the study

Evaluation of ovarian reserve indices in women with normogonadotropic anovulation with SCH and without thyroid disease.

Detailed objectives

i) Assessment of AMH, FSH, LH, estradiol, astral follicle count (AFC)/ovarian volume in the subpopulation of women with PCOS and SCH compared to women with PCOS without thyroid disease ii) Assessment of AMH, FSH, LH, estradiol, AFC/ovarian volume in the subpopulation of women with HPOD (other than PCOS) with SCH compared to women with HPOD without thyroid disease iii) Comparison of AMH, FSH, LH, estradiol, AFC/ovarian volume in women with PCOS and HPOD with and without thyroid disease and evaluation of correlation with US ovarian morphology iv) Calculation of the cut-off point of AMH concentration correlating with a high probability of PCOS diagnosis and TSH correlating with unfavorable parameters of ovarian function/HPO axis.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45
* irregular periods
* infertility due to ovulation disorders
* euthyreosis

Exclusion Criteria:

* diagnosed and treated thyroid dysfunction,
* history of thyroidectomy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study group will consist of women aged 18-45, diagnosed due to menstrual disorders and/or infertility due to ovulation disorders. Inclusion criteria will include age 18-45 and euthyroidism. The exclusion criteria will be: i) diagnosed and treated thyroid dysfunction, ii) history of thyroidectomy. The study population of women will be characterized in terms of demographic (age, BMI) and obstetric data (pregnancy, childbirth, miscarriage, cycle length, infertility).
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Blood serum AMH concentration | 01.07.2022-01.12.2023
  Measurement of serum AMH concentration in women in 4 arms of the study

SECONDARY OUTCOMES:
Blood serum FSH, LH, estradiol | 01.07.2022-01.12.2023
  Measurement of serum FSH, LH, estradiol concentration in women in 4 arms of the study
AFC/ovarian volume | 01.07.2022-01.12.2023
  Ultrasound measurement of AFC/ovarian volume

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jach, Prof., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Department of Gynecology and Obstetrics, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No